CLINICAL TRIAL: NCT01449461
Title: A Phase 1/2 Study of the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of the Oral ALK/EGFR Inhibitor AP26113
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of the Oral Anaplastic Lymphoma Kinase (ALK)/Epidermal Growth Factor Receptor (EGFR) Inhibitor Brigatinib (AP26113)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP26113-11-101; 2011-005718-12 (EudraCT Number); U1111-1196-8197 (Other: World Health Organization)
Record Dates: First submitted 2011-09-30; First posted 2011-10-10 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Lymphoma, Large-Cell, Anaplastic; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Brigatinib 30 mg QD/60 mg QD (Experimental): Brigatinib 30 mg/60 mg, tablets, orally, once daily (QD) in each cycle of 28 days (Approximately up to 7.3 years).
  Interventions: Drug: Brigatinib
- Brigatinib 90 mg QD (Experimental): Brigatinib 90 mg, tablets, orally, QD in each cycle of 28 days (Approximately up to 7.3 years).
  Interventions: Drug: Brigatinib
- Brigatinib 120 mg QD/60 mg BID (Experimental): Brigatinib 120 mg, once daily or 60 mg, twice daily (BID), tablets, orally, in each cycle of 28 days (Approximately up to 7.3 years).
  Interventions: Drug: Brigatinib
- Brigatinib 90 mg QD-180 mg QD (Experimental): Brigatinib 90 mg, tablets, orally, once daily for 7 days followed by brigatinib 180 mg, orally once daily in Cycle 1 of 28 days followed by brigatinib 180 mg, orally once daily in cycle 2 and onward cycles of 28 days.
  Interventions: Drug: Brigatinib
- Brigatinib 180 mg QD/90 mg BID (Experimental): Brigatinib 180 mg, once daily or 90 mg, BID, tablets, orally in each cycle of 28 days (Approximately up to 7.3 years).
  Interventions: Drug: Brigatinib
- Brigatinib 240 mg QD/120 mg BID/300 mg QD (Experimental): Brigatinib 240 mg, QD or 120 mg, BID or 300 mg once daily, tablets, orally, in each cycle of 28 days (Approximately up to 7.3 years).
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib tablets and capsules.
  Other Names: ALUNBRIG™; AP26113

SUMMARY:
The purpose of this study is 2-fold: initially, in the dose escalation phase, the goal is to determine the safety profile of orally administered brigatinib, including: the maximum tolerated dose (MTD), dose limiting toxicities (DLTs), recommended phase 2 dose (RP2D), and pharmacokinetic (PK) profile. Then, once the RP2D is established, an expansion phase will assess the preliminary anti-tumor activity of brigatinib, both in non-small cell lung cancer (NSCLC) with ALK gene rearrangement (including participants with active brain metastases) or mutated EGFR, and in other cancers with abnormal targets against which brigatinib is active.

DETAILED DESCRIPTION:
The drug being tested in this study is called brigatinib (AP26113). Brigatinib is being tested to treat people with NSCLC. This study will look at the safety, tolerability and efficacy of brigatinib.

The study enrolled 137 patients. Participants were assigned to one of the following treatment groups:

* Brigatinib 30 mg once daily (QD)/60 mg QD
* Brigatinib 90 mg QD
* Brigatinib 120 mg QD/60 mg twice daily (BID)
* Brigatinib 90 mg QD-180 mg QD
* Brigatinib 180 mg QD/90 mg BID
* Brigatinib 240 mg QD/120 mg BID/300 mg QD

This multi-center trial will be conducted worldwide. The overall expected time to participate in this study is approximately 4 years. Participants will make multiple visits to the clinic, and 30 days after the End-of-Treatment visit. Follow-up is intended to continue for at least 2 years after the initial dose.

ELIGIBILITY:
Inclusion Criteria:

General Eligibility Criteria

1. All participants must have tumor tissue available for analysis. If sufficient tissue is not available, participants must undergo a biopsy to obtain adequate samples. For participants in expansion cohorts 2, 3 and 5, for whom failure of prior therapy is specified (crizotinib for cohorts 2 and 5, one epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) for cohort 3), tumor tissue must be available following failure of the prior therapy.
2. Must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST).
3. Male or female participants ≥ 18 years old.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Minimum life expectancy of 3 months or more.
6. Adequate renal and hepatic function.
7. Adequate bone marrow function.
8. Normal QT interval on screening electrocardiogram (ECG) evaluation.
9. For females of childbearing potential, a negative pregnancy test must be documented prior to enrollment.
10. Female participants who are of childbearing potential and fertile male participants must agree to use an effective form of contraception with their sexual partners throughout study participation.
11. Signed and dated informed consent indicating that the participant has been informed of all pertinent aspects of the study.
12. Willingness and ability to comply with scheduled visits and study procedures.

Cohort-specific Eligibility Criteria

PART 1: Dose Escalation Phase:

1. Histologically confirmed advanced malignancies. All histologies except leukemia;
2. Refractory to available therapies or for whom no standard or available curative treatments exist;
3. Tumor tissue available for analysis.

PART 2: Expansion cohorts (5 additional cohorts):

1. Expansion cohort 1: Non-small cell lung cancer (NSCLC) participants whose tumors exhibit anaplastic lymphoma kinase (ALK) rearrangements and who have not been treated with previous ALK inhibitors.

i. Histologically or cytologically confirmed NSCLC; ii. Tumor tissue available for analysis (see General Eligibility Criterion 1; iii. History of ALK rearrangement by fluorescence in situ hybridization (FISH); iv. No prior ALK inhibitor therapy; 2. Expansion cohort 2: NSCLC participants whose tumors exhibit ALK rearrangements and who are resistant to crizotinib: i. Histologically or cytologically confirmed NSCLC; ii. Tumor tissue available for analysis (see General Eligibility Criterion 1); iii. History of ALK rearrangement by FISH; iv. Resistant to crizotinib (and have not received any other prior ALK inhibitor therapy); 3. Expansion cohort 3: NSCLC participants whose tumors exhibit an epidermal growth factor receptor EGFR-T790M mutation and who are resistant to 1 prior EGFR TKI: i. Histologically or cytologically confirmed NSCLC ii. Previous treatment with only 1 EGFR TKI for which the last administration was within 30 days of the initiation of brigatinib; iii. Documented evidence of an EGFR-T790M mutation following disease progression on the most recent EGFR TKI therapy; iv. No intervening systemic therapy between cessation of the EGFR TKI and initiating brigatinib; v. Tumor tissue available for analysis (see General Eligibility Criterion 1). 4. Expansion cohort 4: Participants with any cancers with abnormalities in ALK or other brigatinib targets. Examples include, but are not limited to, anaplastic large cell lymphoma (ALCL), diffuse large-cell lymphoma (DLCL), inflammatory myofibroblastic tumors (IMT), and other cancers with ALK abnormalities, or tumors with ROS1 fusions: i. Histologically confirmed lymphomas and other cancers, with the exception of leukemias; ii. Tumor tissue available for analysis (see General Eligibility Criterion 1). 5. Expansion Cohort 5: NSCLC participants whose tumors exhibit ALK rearrangements and who have active, measurable brain metastases: i. Histologically or cytologically confirmed NSCLC: ii. Tumor tissue available for analysis (see General Eligibility Criterion 1); iii. History of ALK rearrangement by FISH; iv. Either crizotinib naive or resistant; v. Have at least one measurable brain lesion (≥ 10 mm by contrast enhanced, T1 weighted magnetic resonance imaging [cMRI]). Previously treated brain lesions by stereotactic radiosurgery (SRS) or surgical resection should not be included as a target or non-target lesion; vi. Previously untreated brain metastases with radiologically documented new or progressing brain lesions. Unequivocal progression of previously treated lesions (non-SRS and non-surgically treated lesions) at least 3 months after the last treatment; vii. Neurologically stable. Participants must be on a stable or deceasing dose of corticosteroids and/or have no requirement for anticonvulsants for 5 days prior to the baseline MRI and for 5 days prior to initiating brigatinib.

Exclusion Criteria:

1. Received an investigational agent ≤ 14 days prior to initiating brigatinib.
2. Received systemic anticancer therapy (including monoclonal antibodies and irreversible TKIs such as afatinib or dacomitinib) or radiation therapy ≤ 14 days prior to initiating brigatinib.

   a. Except for a reversible TKI (ie, erlotinib or gefitinib) or crizotinib, which are allowed up to 72 hours prior to initiating brigatinib, provided that the participant is free of treatment-related toxicity that might confound the safety evaluation of brigatinib.
3. Received any prior agents targeted against ALK, with the exception of crizotinib, or received more than 1 prior EGFR TKI.

   a. Re-challenge with the same TKI is allowed.
4. Major surgery within 28 days prior to initiating brigatinib.
5. Brain metastases that are neurologically unstable or require anticonvulsants or an increasing dose of corticosteroids.

   1. Participants with previously treated brain metastases without evidence of disease or recurrence are allowed for cohorts 1-4.
   2. Participants with evaluable but non-measurable, active brain lesions who otherwise meet the criteria for cohort 5 for CNS disease can be enrolled in other cohorts.
6. Significant uncontrolled or active cardiovascular disease.
7. Uncontrolled hypertension (diastolic blood pressure [BP] > 100 mm Hg; systolic > 150 mm Hg).
8. Prolonged QT interval, or being treated with medications known to cause Torsades de Pointes.
9. History or presence of pulmonary interstitial disease or drug-related pneumonitis.
10. Ongoing or active infection. The requirement for intravenous (IV) antibiotics is considered active infection.
11. Known history of human immunodeficiency virus (HIV). Testing is not required in the absence of history.
12. Pregnant or breastfeeding.
13. Malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of brigatinib.
14. Any condition or illness that, in the opinion of the Investigator, would compromise participant safety or interfere with the evaluation of the safety of the drug.
15. Leptomeningeal carcinomatosis and spinal cord compression. In the case of suspected meningeal involvement, a negative lumbar puncture prior to study entry is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-09-20 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Camidge DR, Kim DW, Tiseo M, Langer CJ, Ahn MJ, Shaw AT, Huber RM, Hochmair MJ, Lee DH, Bazhenova LA, Gold KA, Ou SI, West HL, Reichmann W, Haney J, Clackson T, Kerstein D, Gettinger SN. Exploratory Analysis of Brigatinib Activity in Patients With Anaplastic Lymphoma Kinase-Positive Non-Small-Cell Lung Cancer and Brain Metastases in Two Clinical Trials. J Clin Oncol. 2018 Sep 10;36(26):2693-2701. doi: 10.1200/JCO.2017.77.5841. Epub 2018 May 16. PMID 29768119
- [Derived] Gettinger SN, Bazhenova LA, Langer CJ, Salgia R, Gold KA, Rosell R, Shaw AT, Weiss GJ, Tugnait M, Narasimhan NI, Dorer DJ, Kerstein D, Rivera VM, Clackson T, Haluska FG, Camidge DR. Activity and safety of brigatinib in ALK-rearranged non-small-cell lung cancer and other malignancies: a single-arm, open-label, phase 1/2 trial. Lancet Oncol. 2016 Dec;17(12):1683-1696. doi: 10.1016/S1470-2045(16)30392-8. Epub 2016 Nov 8. PMID 27836716
- [Derived] Yu HA, Riely GJ. Second-generation epidermal growth factor receptor tyrosine kinase inhibitors in lung cancers. J Natl Compr Canc Netw. 2013 Feb 1;11(2):161-9. doi: 10.6004/jnccn.2013.0024. PMID 23411383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in the United States and Spain from 20 September 2011 to 18 February 2020.
Pre-assignment Details: Participants with advanced malignancies, all histologies other than leukemia were enrolled in dose-escalation and participants with non-small cell lung cancer (NSCLC) with anaplastic lymphoma kinase (ALK) rearrangements were enrolled in dose expansion phase. Participants received brigatinib 30 mg - 300 mg, tablets, orally once daily or twice daily.
Groups:
- Brigatinib 90 mg QD-180 mg QD: Brigatinib 90 mg, tablets, orally, once daily for 7 days followed by brigatinib 180 mg, orally QD in Cycle 1 of 28 days followed by brigatinib 180 mg, orally QD in cycle 2 and onward cycles of 28 days (Approximately up to 7.3 years).
Period: Overall Study
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Started | 6 | 18 | 18 | 32 | 48 | 15
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 18 | 18 | 32 | 48 | 15
Not completed — Adverse Event | 0 | 3 | 2 | 3 | 4 | 4
Not completed — Death | 0 | 2 | 0 | 0 | 7 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 4 | 1 | 0
Not completed — Documented Progressive Disease | 4 | 7 | 14 | 15 | 24 | 5
Not completed — Clinical Progressive Disease | 2 | 2 | 0 | 3 | 4 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 1 | 2 | 3 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Reason not Specified | 0 | 1 | 0 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Groups:
- Brigatinib 30 mg QD/60 mg QD: Brigatinib 30 mg/60 mg, tablets, orally, QD in each cycle of 28 days (Approximately up to 7.3 years).
- Brigatinib 120 mg QD/60 mg BID: Brigatinib 120 mg, once daily or 60 mg, BID, tablets, orally, in each cycle of 28 days (Approximately up to 7.3 years).
- Total: Total of all reporting groups
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD | Total
Number analyzed (Participants) | 6 | 18 | 18 | 32 | 48 | 15 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.30) | 57.9 (12.93) | 57.8 (10.91) | 55.7 (11.41) | 53.9 (11.10) | 58.5 (15.60) | 56.4 (12.02)
Age, Customized [Count of Participants; unit: Participants]
  Adults [18-64 years] | 2 | 11 | 12 | 25 | 39 | 9 | 98
  From 65 to 84 years | 4 | 7 | 6 | 7 | 9 | 6 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 13 | 14 | 29 | 8 | 79
  Male | 3 | 6 | 5 | 18 | 19 | 7 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 4 | 3 | 3 | 5 | 2 | 17
  Black or African American | 0 | 1 | 2 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 6 | 13 | 13 | 27 | 39 | 12 | 110
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 5 | 18 | 18 | 31 | 47 | 15 | 134
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 18 | 18 | 32 | 41 | 15 | 130
  Spain | 0 | 0 | 0 | 0 | 7 | 0 | 7
Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — ECOG assessed participant's performance status on a 5 point scale: 0 equals (=) fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, but ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50 percentage [%] of waking hours [h]), capable of all self care, but unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any selfcare, totally confined to bed or chair and 5=Dead.
  Participants
    0 | 0 | 3 | 3 | 13 | 13 | 2 | 34
    1 | 6 | 15 | 15 | 19 | 33 | 13 | 101
    2 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Time Since Diagnosis of Cancer [Mean (Standard Deviation); unit: years] | 2.48 (3.303) | 3.33 (2.184) | 2.41 (1.346) | 3.19 (2.726) | 2.77 (2.053) | 3.27 (1.913) | 2.93 (2.192)
Participants with Diagnosis of Cancer Type [Count of Participants; unit: Participants]
  NSCLC | 3 | 16 | 18 | 31 | 45 | 15 | 128
  Other | 3 | 2 | 0 | 1 | 3 | 0 | 9
Number of Participants with Mutation Types [Count of Participants; unit: Participants]
  Anaplastic Lymphoma Kinase (ALK+) | 1 | 16 | 6 | 29 | 27 | 5 | 84
  Epidermal Growth Factor Receptor (EGFRm) | 2 | 1 | 10 | 3 | 18 | 9 | 43
  ROS Proto-oncogene 1 (ROS1+) | 0 | 0 | 0 | 0 | 3 | 1 | 4
  Other | 3 | 1 | 2 | 0 | 0 | 0 | 6
Participants with Prior Chemotherapy Regimen [Count of Participants; unit: Participants]
  0 | 0 | 2 | 7 | 12 | 12 | 3 | 36
  1 | 3 | 4 | 3 | 6 | 17 | 2 | 35
  2 | 0 | 9 | 4 | 8 | 10 | 5 | 36
  > 2 | 3 | 3 | 4 | 6 | 9 | 5 | 30
Participants with Prior Radiotherapy to Brain [Count of Participants; unit: Participants]
  No | 6 | 13 | 17 | 24 | 36 | 14 | 110
  Yes | 0 | 5 | 1 | 8 | 12 | 1 | 27

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Brigatinib
Description: The RP2D is the maximum tolerated dose (MTD) or less. The MTD is defined as the dose range at which ≤ 1 of 6 evaluable participants experience dose limiting toxicities (DLT) within the first 28 days of treatment (end of Cycle 1).
Time Frame: 28 days
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Mean (Full Range); unit: mg
Groups:
- Brigatinib: All participants who received brigatinib, tablets, orally, once daily in each cycle of 28 days (Approximately up to 7.3 years).
Arm/Group | Brigatinib
Number analyzed (Participants) | 137
mg | NA [90 to 180] — RP2D for this study is a dose range.

2. Primary Outcome: Objective Response Rate (ORR)
Description: ORR assessed by the investigator, is defined as the percentage of the participants with complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid tumors (RECIST) v1.1 after the initiation of study treatment. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: Disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and normalization of tumor marker level. PR: at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline sum diameters. Crzb=Crizotinib.
Time Frame: From Screening and at 8-week intervals thereafter up to end of the study (up to 8.4 years)
Population: Full analysis set (FAS) included all participants who received at least one dose of study drug. Participants with anaplastic lymphoma kinase (ALK) and non-small cell lung cancer (NSCLC) were evaluated for this outcome measure. Number analyzed is the number of participants with data evaluable for specific category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 1 | 14 | 6 | 28 | 25 | 5
percentage of participants
  With Prior Treatment with Crizotinib: number analyzed (Participants) | 1 | 13 | 5 | 25 | 23 | 4
  With Prior Treatment with Crizotinib | 0 [0 to 0] | 53.8 [25.1 to 80.8] | 60.0 [14.7 to 94.7] | 76.0 [54.9 to 90.6] | 65.2 [42.7 to 83.6] | 25.0 [0.6 to 80.6]
  Without Prior Treatment with Crizotinib: number analyzed (Participants) | 0 | 1 | 1 | 3 | 2 | 1
  Without Prior Treatment with Crizotinib |  | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [2.5 to 100.0]

3. Secondary Outcome: Number of Participants Who Had at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug up to 30 days following the last dose of the study treatment or the investigator/participant decision to discontinue treatment, whichever occurs first (approximately up to 7.4 years)
Population: Safety population included all enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 6 | 18 | 18 | 32 | 48 | 15
Participants | 6 | 18 | 18 | 32 | 48 | 15

4. Secondary Outcome: Maximum Tolerated Dose (MTD) Assessed in Dose Escalation Phase of the Study
Description: The MTD is defined as the highest dose at which ≤ 1 of 6 evaluable participants experience a DLT within the first 28 days of treatment (end of Cycle 1).
Time Frame: Up to Cycle 1 (28 days)
Population: Safety population included all enrolled participants who received at least one dose of study drug. Participants enrolled in the dose escalation phase were included in the analysis.
Measure: Number; unit: mg
Groups:
- Brigatinib: All participants received brigatinib tablets, orally, once daily (QD) starting at 30 mg in each cycle of 28 days.
Arm/Group | Brigatinib
Number analyzed (Participants) | 66
mg | NA — MTD criteria was not met.

5. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Assessed in Dose Escalation Phase of the Study
Description: DLT include any toxicity that is possibly, probably, or definitely drug-related. Toxicity grades will be defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.0. DLTs are defined by the following: A) Non-hematologic toxicities: Any grade ≥3 non-hematologic toxicity, with the exception of self-limiting or medically controllable toxicities (eg, nausea, vomiting, fatigue, electrolyte disturbances, hypersensitivity reactions) lasting < 3 days, and excluding alopecia. B) Hematologic toxicities: Febrile neutropenia not related to underlying disease (fever, > 101°F; ANC<500); Prolonged grade 4 neutropenia (> 7 days); Neutropenic infection: ≥ grade 3 neutropenia with ≥ grade 3 infection; Thrombocytopenia ≥ grade 3 with bleeding or grade 4 lasting ≥ 7 days. C) Missed ≥ 25% of planned doses of brigatinib over 28 days due to treatment-related AEs in the first cycle.
Time Frame: Up to Cycle 1 (28 days)
Population: DLT-evaluable population included participants who received ≥75% of planned study drug doses during Cycle 1.
Measure: Number; unit: participants
Groups:
- Brigatinib 30 mg: Brigatinib 30 mg, tablets, orally, once daily (QD) in each cycle of 28 days (Approximately up to 7.3 years).
- Brigatinib 60 mg: Brigatinib 60 mg, tablets, orally, once daily (QD) in each cycle of 28 days (Approximately up to 7.3 years).
- Brigatinib 90 mg: Brigatinib 90 mg, tablets, orally, once daily or twice daily in each cycle of 28 days (Approximately up to 7.3 years).
- Brigatinib 120 mg: Brigatinib 120 mg, tablets, orally, once daily in each cycle of 28 days (Approximately up to 7.3 years).
- Brigatinib 180 mg: Brigatinib 180 mg, tablets, orally once daily in each cycle of 28 days (Approximately up to 7.3 years).
- Brigatinib 240 mg: Brigatinib 240 mg, tablets, orally, once daily in each cycle of 28 days (Approximately up to 7.3 years).
- Brigatinib 300 mg: Brigatinib 300 mg, tablets, orally, once daily in each cycle of 28 days (Approximately up to 7.3 years).
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 6 | 2
participants | 0 | 0 | 0 | 0 | 0 | 1 | 1

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Brigatinib at Cycle 1 Day 1
Time Frame: Cycle 1 (28-days cycle): Day 1
Population: Analysis was performed on all enrolled participants in the study who received at least one dose of brigatinib. Here number of participants analyzed is the participants who were evaluable for this outcome measure. Participants of brigatinib 90 mg QD-180 mg QD arm were included as per treatment received at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 3 | 3 | 50 | 11 | 44 | 10 | 2
ng/mL | 125.6 (41.07) | 406.3 (102) | 493 (289.5) | 793.7 (828.7) | 1185 (607.6) | 1515 (637.9) | 895 (487.9)

7. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Brigatinib at Cycle 2 Day 1
Time Frame: Cycle 2 (28-days cycle): Day 1
Population: Analysis was performed on all enrolled participants in the study who received at least one dose of brigatinib. Here number of participants analyzed is the participants with data available for analysis for this outcome measure. Participants of brigatinib 90 mg QD-180 mg QD arm were included as per treatment received at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 2 | 3 | 15 | 10 | 63 | 7 | 0
ng/mL | 249.50 (167.58) | 491.67 (223.95) | 634.07 (310.05) | 942.30 (472.33) | 1694.3 (1014.3) | 2280.0 (1308.5) |

8. Secondary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for Brigatinib at Cycle 1 Day 1
Time Frame: Cycle 1 (28-days cycle): Day 1
Population: Analysis was performed on all enrolled participants in the study who received at least one dose of brigatinib. Here, number of participants analyzed is the participants who were evaluable for this outcome measure. Participants of brigatinib 90 mg QD-180 mg QD arm were included as per treatment received at each time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 3 | 3 | 50 | 11 | 44 | 10 | 2
hours | 3.9 [3.8 to 4.0] | 1.0 [0.48 to 4.0] | 2.0 [0.48 to 24] | 2.0 [0.98 to 6.0] | 2.0 [0.60 to 25] | 2.0 [1.0 to 4.0] | 4.05 [4 to 4.1]

9. Secondary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for Brigatinib at Cycle 2 Day 1
Time Frame: Cycle 2 (28-days cycle): Day 1
Population: Analysis was performed on all enrolled participants in the study who received at least one dose of brigatinib. Here, number of participants analyzed is the participants with data available for analyses for this outcome measure. Participants of brigatinib 90 mg QD-180 mg QD arm were included as per treatment received at each time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 2 | 3 | 15 | 10 | 63 | 7 | 0
hours | 2.49 [0.98 to 4.0] | 1.00 [0.50 to 1.8] | 2.00 [0.98 to 8.0] | 3.00 [0.50 to 6.1] | 2.10 [0.50 to 6.2] | 2.00 [1.0 to 4.0] |

10. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Post-dose for Brigatinib at Cycle 1 Day 1
Time Frame: Cycle 1 (28-days cycle): Day 1 multiple time points (up to 24 hours) post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 3 | 3 | 15 | 11 | 63 | 7 | 2
h*ng/mL | 1320.9 (576.29) | 3900 (430.31) | 5710.1 (3268.4) | 9895.5 (11772) | 13204 (6306.9) | 16800 (7571.1) | 12356 (5869)

11. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Post-dose for Brigatinib at Cycle 2 Day 1
Time Frame: Cycle 2 (28-days cycle): Day 1 multiple time points (up to 24 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 2 | 3 | 15 | 10 | 63 | 7 | 0
h*ng/mL | 2689.0 (1145.5) | 5069.0 (1664.7) | 9142.1 (4076.7) | 13888 (7011.4) | 23478 (14463) | 30117 (19921) |

12. Secondary Outcome: T1/2: Terminal Phase Elimination Half-life for Brigatinib at Cycle 2 Day 1
Time Frame: Cycle 2 (28-days cycle): Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Brigatinib 30 mg | Brigatinib 60 mg | Brigatinib 90 mg | Brigatinib 120 mg | Brigatinib 180 mg | Brigatinib 240 mg | Brigatinib 300 mg
Number analyzed (Participants) | 2 | 3 | 15 | 10 | 63 | 7 | 0
hours | 31.55 (2.758) | 30.93 (5.873) | 28.69 (10.06) | 25.52 (7.958) | 24.90 (7.437) | 21.77 (4.007) |

13. Secondary Outcome: Best Overall Response
Description: Best overall response is defined as percentage of participants with CR, PR, stable disease (SD) or progressive disease (PD) as per of RECIST v1.1 as evaluated by investigator. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and normalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters. Disease progression for target lesion: SLD increased by at least 20% from smallest value on study and SLD must also demonstrate an absolute increase of at least 5 mm or development of any new lesion. PD for non-target lesion: unequivocal progression of existing non-target lesions. SD for neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Screening and at 8-week intervals thereafter up to end of the study (up to 8.4 years)
Population: Full analysis set included all participants who received at least one dose of study drug. Participants with ALK and NSCLC were evaluated for this outcome measure. Number analyzed is the number of participants with data evaluable for specific category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 1 | 14 | 6 | 28 | 25 | 5
percentage of participants
  With Prior Treatment with Crizotinib: Complete Response: number analyzed (Participants) | 1 | 13 | 5 | 25 | 23 | 4
  With Prior Treatment with Crizotinib: Complete Response | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 12.0 [2.5 to 31.2] | 8.7 [1.1 to 28.0] | 0.0 [0.0 to 0.0]
  Without Prior Treatment with Crizotinib: Complete Response: number analyzed (Participants) | 0 | 1 | 1 | 3 | 2 | 1
  Without Prior Treatment with Crizotinib: Complete Response |  | 0.0 [0.0 to 0.0] | 100.0 [2.5 to 100.0] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 0.0] | 100.0 [2.5 to 100.0]
  With Prior Treatment with Crizotinib: Partial Response: number analyzed (Participants) | 1 | 13 | 5 | 25 | 23 | 4
  With Prior Treatment with Crizotinib: Partial Response | 0.0 [0.0 to 0.0] | 53.8 [25.1 to 80.8] | 60.0 [14.7 to 94.7] | 64.0 [42.5 to 82.0] | 56.5 [34.5 to 76.8] | 25.0 [0.6 to 80.6]
  Without Prior Treatment with Crizotinib: Partial Response: number analyzed (Participants) | 0 | 1 | 1 | 3 | 2 | 1
  Without Prior Treatment with Crizotinib: Partial Response |  | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 0.0] | 66.7 [9.4 to 99.2] | 100.0 [15.8 to 100.0] | 0.0 [0.0 to 0.0]
  With Prior Treatment with Crizotinib: Stable Disease: number analyzed (Participants) | 1 | 13 | 5 | 25 | 23 | 4
  With Prior Treatment with Crizotinib: Stable Disease | 100.0 [2.5 to 100.0] | 23.1 [5.0 to 53.8] | 0.0 [0.0 to 0.0] | 12.0 [2.5 to 31.2] | 13.0 [2.8 to 33.6] | 75.0 [19.4 to 99.4]
  Without Prior Treatment with Crizotinib: Stable Disease: number analyzed (Participants) | 0 | 1 | 1 | 3 | 2 | 1
  Without Prior Treatment with Crizotinib: Stable Disease |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  With Prior Treatment with Crizotinib: Progressive Disease: number analyzed (Participants) | 1 | 13 | 5 | 25 | 23 | 4
  With Prior Treatment with Crizotinib: Progressive Disease | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 8.0 [1.0 to 26.0] | 21.7 [7.5 to 43.7] | 0.0 [0.0 to 0.0]
  Without Prior Treatment with Crizotinib: Progressive Disease: number analyzed (Participants) | 0 | 1 | 1 | 3 | 2 | 1
  Without Prior Treatment with Crizotinib: Progressive Disease |  | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

14. Secondary Outcome: Duration of Response
Description: Duration of response is defined as time interval from time that measurement criteria are first met for CR/PR (whichever is first recorded) until first date that progressive disease is objectively documented or death due to any cause. Participants who did not progress nor die were censored at last valid response assessment.CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis.CR for non-target lesion:disappearance of all extranodal non-target lesions,all lymph nodes must be non-pathological in size(<10mm short axis) and normalization of tumor marker level.PR:at least a 30% decrease in SLD of target lesions.PD for target lesion:SLD increased by at least 20% from smallest value and must also demonstrate an absolute increase of >=5 mm or development of any new lesion.PD for non-target lesion:unequivocal progression of existing non-target lesions.Duration of response calculated by Kaplan-Meier estimation.
Time Frame: Screening and at 8-week intervals thereafter up to end of the study (up to 8.4 years)
Population: Full analysis set included all participants who received at least one dose of study drug. Participants who were responders among those who had ALK and NSCLC were evaluated for this outcome measure. Number analyzed is the number of participants with data evaluable for specific category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 0 | 8 | 4 | 22 | 17 | 2
months
  With Prior Treatment with Crizotinib: number analyzed (Participants) | 0 | 7 | 3 | 19 | 15 | 1
  With Prior Treatment with Crizotinib |  | 11.1 [3.8 to 16.7] | 4.0 [3.7 to 29.5] | 14.8 [7.9 to 25.1] | 20.4 [7.5 to 51.6] | 29.7 [NA to NA] — 95% CI was not estimable due to low number of participants with events.
  Without Prior Treatment with Crizotinib: number analyzed (Participants) | 0 | 1 | 1 | 3 | 2 | 1
  Without Prior Treatment with Crizotinib |  | 30.4 [NA to NA] — 95% CI was not estimable due to low number of participants with events. | 60.3 [NA to NA] — 95% CI was not estimable due to low number of participants with events. | 52.0 [5.6 to 52.0] | 20.8 [9.2 to 32.4] | NA [NA to NA] — Duration of response was not estimable due to low number of participants with events.

15. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time interval from the date of the first dose of the study treatment until the first date at which disease progression is objectively documented, or death due to any cause, whichever occurs first. Disease progression for target lesion: SLD increased by at least 20% from the smallest value on study (including baseline, if that is the smallest) and SLD must also demonstrate an absolute increase of at least 5 mm or development of any new lesion. Disease progression for non-target lesion: Unequivocal progression of existing non-target lesions. (Subjective judgment by experienced reader).
Time Frame: Screening and at 8-week intervals thereafter up to end of the study (up to 8.4 years)
Population: Analysis was performed on all enrolled participants in the study who received at least one dose of brigatinib. Here, overall number of participants analyzed is the participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 5 | 15 | 17 | 21 | 40 | 7
months | 1.8 [1.0 to 5.5] | 12.6 [0.9 to 47.9] | 5.4 [0.8 to 63.9] | 11.0 [0.5 to 53.6] | 5.4 [0.1 to 69.9] | 5.4 [1.8 to 31.5]

16. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval from the date of the first dose of the study treatment until death due to any cause.
Time Frame: Screening and at 8-week intervals thereafter up to end of the study (up to 8.4 years)
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 6 | 11 | 12 | 17 | 25 | 11
months | 5.3 [2.3 to 12.6] | 11.6 [4.0 to 47.6] | 7.3 [0.5 to 28.6] | 17.9 [1.4 to 35.0] | 7.3 [0.1 to 55.0] | 8.3 [3.3 to 22.3]

17. Secondary Outcome: Intracranial Objective Response Rate
Description: Intracranial objective response rate is defined as the percentage of the participants with CR or PR in the intracranial CNS per modification of RECIST v1.1 after the initiation of study drug. CR for target lesion: disappearance of all extranodal lesions. CR for non-target lesion: disappearance of all extranodal non-target lesions and normalization of tumor marker level. PR: at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline sum diameters.
Time Frame: Screening and at 8-week intervals thereafter (approximately up to 50 months)
Population: Full analysis set. ALK+ NSCLC participants with measurable and non-measurable brain metastases at baseline were evaluated for this outcome measure. Here, number analyzed is the number of participants who were evaluable for specific category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 0 | 8 | 1 | 18 | 16 | 3
percentage of participants
  Measurable Brain Metastases: number analyzed (Participants) | 0 | 2 | 0 | 5 | 7 | 1
  Measurable Brain Metastases |  | 100 [15.8 to 100] |  | 80 [28.4 to 99.5] | 42.9 [9.9 to 81.6] | 100 [2.5 to 100]
  Only Non-Measurable Brain Metastases: number analyzed (Participants) | 0 | 6 | 1 | 13 | 9 | 2
  Only Non-Measurable Brain Metastases |  | 16.7 [0.4 to 64.1] | 100 [2.5 to 100] | 46.2 [19.2 to 74.9] | 44.4 [13.7 to 78.8] | 50.0 [1.3 to 98.7]

18. Secondary Outcome: Duration of Intracranial Response
Description: Intracranial duration of response is defined as the time interval from the time that the measurement criteria are first met for CR/PR in brain metastases (whichever is first recorded) until the first date that progressive disease is objectively documented or death due to any cause. Participants who did not progress nor die were censored at the last valid response assessment. Duration intracranial of response was calculated by Kaplan-Meier estimation.
Time Frame: Screening and at 8-week intervals thereafter (approximately up to 50 months)
Population: Full analysis set. ALK+ NSCLC participants with measurable and non-measurable brain metastases at baseline were evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 0 | 8 | 1 | 18 | 16 | 3
months |  | 12.9 [NA to NA] — Upper and lower limit of duration of intracranial response was not reached due to low number of participants with events. | 5.0 [NA to NA] — Upper and lower limit of duration of intracranial response was not reached due to low number of participants with events. | 11.4 [7.5 to 11.4] | 29.2 [5.5 to 29.2] | 11.3 [3.6 to 18.9]

19. Secondary Outcome: Intracranial Progression Free Survival (PFS)
Description: PFS is defined as the time interval from the date of the first dose of the study treatment until the first date at which disease progression in brain, or death due to any cause, whichever occurs first. Intracranial PFS was calculated by Kaplan-Meier estimation.
Time Frame: Screening and at 8-week intervals thereafter (approximately up to 50 months)
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
Number analyzed (Participants) | 0 | 8 | 1 | 18 | 16 | 3
months |  | 36.8 [5.5 to 36.8] | 6.7 [NA to NA] — Upper limit of 95% CI was not reached due to low number of participants with events. | NA [9.4 to NA] — Progression-free survival was not reached due to low number of participants with events. | 14.4 [7.3 to 31.1] | 7.3 [3.1 to 22.3]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From first dose up to the End of the Study (Up to 8.4 years). Serious and other adverse events: From first dose of study drug up to 30 days following the last dose of the study treatment or the investigator/participant decision to discontinue treatment, whichever occurs first (approximately up to 7.4 years)
Arm/Group | Brigatinib 30 mg QD/60 mg QD | Brigatinib 90 mg QD | Brigatinib 120 mg QD/60 mg BID | Brigatinib 90 mg QD-180 mg QD | Brigatinib 180 mg QD/90 mg BID | Brigatinib 240 mg QD/120 mg BID/300 mg QD
All-Cause Mortality (participants affected / at risk) | 6/6 | 11/18 | 12/18 | 17/32 | 25/48 | 11/15
Serious Adverse Events (participants affected / at risk) | 1/6 | 10/18 | 10/18 | 14/32 | 30/48 | 11/15
Other Adverse Events (participants affected / at risk) | 6/6 | 17/18 | 17/18 | 31/32 | 45/48 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 30 mg QD/60 mg QD (N=6) | Brigatinib 90 mg QD (N=18) | Brigatinib 120 mg QD/60 mg BID (N=18) | Brigatinib 90 mg QD-180 mg QD (N=32) | Brigatinib 180 mg QD/90 mg BID (N=48) | Brigatinib 240 mg QD/120 mg BID/300 mg QD (N=15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 3 | 1 | 4 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 1 | 1 | 5 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bezoar (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal compression (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Radiation associated cardiac failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 30 mg QD/60 mg QD (N=6) | Brigatinib 90 mg QD (N=18) | Brigatinib 120 mg QD/60 mg BID (N=18) | Brigatinib 90 mg QD-180 mg QD (N=32) | Brigatinib 180 mg QD/90 mg BID (N=48) | Brigatinib 240 mg QD/120 mg BID/300 mg QD (N=15)
Nausea (Gastrointestinal disorders) | 3 | 8 | 9 | 16 | 33 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 7 | 17 | 21 | 8
Constipation (Gastrointestinal disorders) | 1 | 6 | 5 | 9 | 8 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 5 | 9 | 19 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2 | 6 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 5 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 4 | 1 | 1 | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 5 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 1 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 3
Aphthous ulcer (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 6 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal irritation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 2 | 9 | 9 | 16 | 19 | 12
Oedema peripheral (General disorders) | 1 | 1 | 4 | 6 | 5 | 4
Pyrexia (General disorders) | 0 | 3 | 2 | 6 | 7 | 2
Pain (General disorders) | 0 | 3 | 2 | 4 | 3 | 1
Chest discomfort (General disorders) | 0 | 3 | 0 | 3 | 5 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 2 | 1 | 3 | 3
Influenza like illness (General disorders) | 0 | 1 | 2 | 4 | 3 | 1
Asthenia (General disorders) | 0 | 1 | 1 | 1 | 5 | 1
Chills (General disorders) | 0 | 3 | 0 | 3 | 2 | 2
Gait disturbance (General disorders) | 0 | 1 | 0 | 2 | 4 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0 | 2 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 2 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Exercise tolerance decreased (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Feeling jittery (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 6 | 13 | 14 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 5 | 7 | 10 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 5 | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 4 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 4 | 5 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 0 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 4 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 3 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 3 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 2 | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 1 | 0 | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 5 | 4 | 3
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Radiation neuropathy (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 4 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 6 | 11 | 10 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vascular pain (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 6 | 6 | 3
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 5 | 2 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 4 | 3 | 0
Bruxism (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Anticipatory anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 2 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 2 | 6 | 5 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 1
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0
Photopsia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 12 | 7 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1 | 4 | 5 | 7 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 6 | 9 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 4 | 3 | 4
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 2 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 3 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasal herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3 | 3 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 3 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 7 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 4 | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 4 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 5 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 3 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5 | 1 | 10 | 12 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 7 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 4 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 5 | 5 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 5 | 5 | 10 | 9 | 3
Lipase increased (Investigations) | 0 | 5 | 4 | 12 | 6 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 7 | 10 | 9 | 2
Alanine aminotransferase increased (Investigations) | 0 | 3 | 3 | 6 | 5 | 1
Blood insulin increased (Investigations) | 0 | 4 | 2 | 4 | 5 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 5 | 6 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 2 | 4 | 4 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 2 | 2 | 1
Weight increased (Investigations) | 0 | 1 | 2 | 1 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 1 | 2 | 1
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 2 | 4 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 2 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1 | 1 | 3 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 1 | 0 | 1 | 2 | 1
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Urinary sediment present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 8 | 13 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5 | 11 | 10 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3 | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 10 | 10 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 2 | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 4 | 3 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 5 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 6 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 6 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 8 | 7 | 14 | 18 | 6
Dizziness (Nervous system disorders) | 0 | 5 | 1 | 5 | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 2 | 6 | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 1 | 2 | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1 | 3 | 3 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 2 | 3 | 0
Balance disorder (Nervous system disorders) | 0 | 2 | 0 | 2 | 5 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 4 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 5 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 2
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1 | 3 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 2 | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 2 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 2 | 1 | 1 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 2 | 4 | 3 | 1
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood sodium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Ear infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 2 | 2 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dyschromatopsia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cataract cortical (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased. (Investigations) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT01449461/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT01449461/SAP_001.pdf